CLINICAL TRIAL: NCT02257164
Title: Anesthesic Techniques for Surgery of the Anterior Cruciate Ligament of the Knee in Ambulatory Surgery. Randomized Pilot Monocentric Trial
Acronym: CLICA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1408021; 2014-002062-77 (EudraCT Number)
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: anterior cruciate ligament reconstruction; femoral nerve block; articular injection and obturator nerve block
MeSH Terms: interventions — Injections, Intra-Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- femoral nerve block (Active Comparator): 20 ml injection of 2 mg/ml ropivacaine in femoral nerve
  Interventions: Procedure: Femoral nerve block
- obturator nerve block and intraarticular injection (Experimental): 10 ml injection of 2 mg/ml ropivacaine in obturator nerve intraarticular injection : 10 ml of chlorhydrate ropivacaine (2 mg/ml) and 10ml of magnesium sulfate
  Interventions: Procedure: obturator nerve block; Procedure: intraarticular injection

INTERVENTIONS:
Procedure: Femoral nerve block — 2 mg/ml
  Arms: femoral nerve block
Procedure: obturator nerve block
  Arms: obturator nerve block and intraarticular injection
Procedure: intraarticular injection
  Arms: obturator nerve block and intraarticular injection

SUMMARY:
Surgery of the anterior cruciate ligament of the knee is frequently a young patient surgery. The post-operative pain of this surgery is managed according to recommendation. In the majority of case, femoral nerve block is performed. The femoral nerve block can cause "paralysis" of the quadriceps more or less complete that no allowing a good quadriceps locking. This locking is indispensable to avoid post-operative flexima and to ensure stabilization of the knee during walking.

In France, the surgery requires a duration of hospitalization from 2 to 4 days in the most cases. It is sometimes performed in ambulatory especially in the USA. But, at the home, pain requires powerful analgesics with their adverse events.

Today, no anesthesic technics for surgery of anterior cruciate ligament of the knee ensure in the same time optimal analgesia and optimal quadriceps locking. The main objective of the investigators study is to compare two analgesia techniques : femoral nerve block vs intra articular injection and obturator nerve block in surgery of the anterior cruciate ligament of the knee

ELIGIBILITY:
Inclusion Criteria:

* Physical Status score = 1 or Physical Status score = 2
* Major Patient
* indication of anterior cruciate ligament reconstruction
* informed consent for participation in the study

Exclusion Criteria:

* Contraindication to general analgesia
* Contraindication to peripheral nerve block
* Allergy to analgesic treatment
* Porphyria,
* Neurologic deficit
* Contraindication antiinflammatory drugs
* Simultaneous reconstruction of another ligament or complex gesture intended
* Patient treated with an anti-arrhythmic drug class III
* Patient with severe hepatic impairment
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
number of patients with success | 4 postoperative hours
  success is defined by : score chung > or egal to 9 and quadriceps locking > or egal to 3/5

SECONDARY OUTCOMES:
Pain for all patients | Postoperative hours : 0, 1, 2, 4, 6, 8, 12, 18, 24, 36 and 48
  pain measured by EVA
analgesic consumption for all patients | Postoperative hours : 0, 1, 2, 4, 6, 8, 12, 18, 24, 36 and 48
  analgesic consumption of tramadol and morphine (use, number)
analgesic adverse events for all patients | Postoperative hours : 0, 1, 2, 4, 6, 8, 12, 18, 24, 36 and 48
  Frequency of nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie PASSOT, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- PASSOT, Saint-Etienne, France